CLINICAL TRIAL: NCT04635553
Title: Prevalence of Potential Schistosome Hybrids and Their Invasive Capacity Under Praziquantel Pressure in Northern Senegal
Brief Title: Monitoring Schistosome Hybrids Under Under Praziquantel Pressure
Acronym: Sen_hybrids
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Sponsor
Other Study IDs: SEN2020-BS
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-09

CONDITIONS: Schistosomiasis
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Schistosome miracidia
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Praziquantel 600 milligram — A single treatment with a dose of 40 milligram/kilogram (mg/kg)

SUMMARY:
The overall objective of this project is to examine and quantify the potential existence and impact on Praziquantel (PZQ) efficacy, of naturally occurring S. haematobium and S. bovis hybrid populations in northern Senegal. Schistosome hybrids may present vigor compared to their pure parental forms and hence, may be less sensitive to PZQ. We hypothesise that PZQ repeated treatment selects the hybrid schistosome populations.

DETAILED DESCRIPTION:
Human schistosomiasis is a Neglected Tropical Disease caused by schistosome helminth worms with impressive epidemiological statistics associated: 800 million people at risk in 78 countries, > 230 million infected and > 200 000 deaths each year. The disease is highly endemic in sub-Saharan Africa where it persists despite mass drug administration with Praziquantel (PZQ). Some schistosomes are specific to humans and induce two main disease forms (either mesenteric or uro-genital) while others are associated with wild animals. However, hybridization can occur between different schistosome species. In northern Senegal, hybridization between schistosome species specific to humans and animals is now known to be frequent with the potential risk of zoonotic transmission.

This study will propose an integrative approach by conducting parasitological and molecular analysis including, schistosome miracidia genotyping to show if PZQ repeated treatment affects the genomic composition (Frequencies of alleles) of hybrid populations.

The objectives are:

* Determine the current prevalence of potential hybrid schistosome populations in their natural setting in Senegal
* Determine the sensitivity of hybrid schistosomes to praziquantel treatment in field populations
* Determine the molecular basis (at the genome level) of such phenotypic changes).

The study is a longitudinal observation of a cohort of school children after repeated Praziquantel (40 mg/kg) treatment, a drug commonly used through Mass Drug Administration (MDA) to treat schistosomiasis.

The cohort will be followed over a period of three years. Before the followup, a baseline urogenital schistosomiasis test will be performed on 1, 450 school-age children randomly selected in the five sites (290 in each site). All positive children will receive a single treatment (T1) of Praziquantel (PZQ) (40 mg/kg). Among those who test positive for S. haematobium eggs, only 50 in each site (five sites), who meet all the eligibility criteria will be invited to participate to the longitudinal follow-up. Four rounds of a single praziquantel (PZQ) treatment will be administered to positive individuals every 6 months. One round will consist of one treatment (T1 to T4) followed by a control treatment after one month (CT1 to CT4), hence, before the potential re-infecting schistosomes become adults and start egg-laying, which could bias the effectiveness of treatment evaluations. At each CT time, samples will be collected and S. haematobium eggs quantified (number of excreted eggs/10 mls of urine). Parasites (miracidia hatched from excreted eggs) will be recovered before each initial treatment (T1 to T4) and at CT1 to CT4 for subsequent genetic analysis to characterize hybrid schistosomes between S. haematobium and S. bovis.

ELIGIBILITY:
Inclusion Criteria:

* Children between the initiation courses (CI) and elementary course second year (CE2)
* Absence of declared chronic pathologies that could impact the follow-up
* Be positive for S. haematobium infection during the selection period (excreting eggs)
* Residing in the study area during the 3 years of the follow-up

Exclusion Criteria:

* Absence of written informed consent or expressed refusal from the child
* Enrolled in another on going study, which implicates the administration of PZQ or tests another product.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Northern Senegal Children
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in prevalence and intensity of schistosome infection | December 31. 2020
  Determine at the 1 month post treatment the cure rate (CR) of the treatments and Egg Reduction Rates (ERR).

SECONDARY OUTCOMES:
Hybrids tolerance to praziquantel | December 31, 2021
  The frequency of hybrids and the level of genomic introgression between S. bovis and S. haematobium

CONTACTS AND LOCATIONS:
Locations (1):
- Bruno SENGHOR, Dakar, Senegal

REFERENCES:
- [Derived] Senghor B, Mathieu-Begne E, Rey O, Doucoure S, Sow D, Diop B, Sene M, Boissier J, Sokhna C. Urogenital schistosomiasis in three different water access in the Senegal river basin: prevalence and monitoring praziquantel efficacy and re-infection levels. BMC Infect Dis. 2022 Dec 29;22(1):968. doi: 10.1186/s12879-022-07813-5. PMID 36581796